CLINICAL TRIAL: NCT00542126
Title: Luteal-Phase GnRH Agonist Administration in Frozen-Thawed IVF Embryo Transfer Cycles
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GnRHFETsupport.CTIL
Record Dates: First submitted 2007-09-19; First posted 2007-10-10 (Estimated); Last update posted 2007-10-10 (Estimated); Status verified 2007-09

CONDITIONS: Pregnancy Rate
Keywords: GnRH analog, IVF, infertility, frozen-thawed embryos
MeSH Terms: conditions — Infertility | interventions — Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): GnRH analog administration following embryo transfer
  Interventions: Drug: Decapeptyl 0.1 mg after embryo transfer
- 2 (No Intervention)

INTERVENTIONS:
Drug: Decapeptyl 0.1 mg after embryo transfer — Decapeptyl 0.1 mg (Ferring, Kiel, Germany) 3 days following embryo transfer
  Arms: 1

SUMMARY:
Supraphysiological hormonal stimulation enables collecting many oocytes in an In-Vitro Fertilization treatment, but may have a negative effect on uterine function and contribute the fact that the majority of preembryos placed in the uterus fail to implant.

Several medical agents were shown to be beneficial when given in the luteal phase of an IVF cycle, but the optimal regimen has not been yet determined. In 2006, a European group reported that addition of GnRH analog (Decapeptyl) as luteal support in IVF cycle significantly improved pregnancy and delivery rates. It is not known whether this positive effect influences the corpus luteum, embryo or the uterus. The researchers sought to evaluate the effect of GnRH administration as luteal support in frozen-thaws IVF cycle.

ELIGIBILITY:
Inclusion Criteria:

IVF patients transfer of a minimum of two medium-quality thawed embryos in IVF

Exclusion Criteria:

1. Two or more fresh IVF embryo transfer or three or more thawed embryos transfer with no pregnancy.
2. maximal endometrial thickness < 6 mm or intracavitary fluid at the time of embryo transfer on previous cycles
3. Untreated hydrosalpinges
4. intracavitary mass
5. submucous myoma
6. known allergy to one of medical agents used in the study

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2007-12; Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
pregnancy and delivery rates

CONTACTS AND LOCATIONS:
Overall Officials: Avi Tsafrir, MD, Principal Investigator — Shaare-Zedek Medical Center, Jerusalem, Israel
Locations (1):
- IVF unit, Shaare-Zedek Medical Center, Jerusalem, Israel

REFERENCES:
- [Background] Tesarik J, Hazout A, Mendoza-Tesarik R, Mendoza N, Mendoza C. Beneficial effect of luteal-phase GnRH agonist administration on embryo implantation after ICSI in both GnRH agonist- and antagonist-treated ovarian stimulation cycles. Hum Reprod. 2006 Oct;21(10):2572-9. doi: 10.1093/humrep/del173. Epub 2006 Aug 22. PMID 16926261